CLINICAL TRIAL: NCT00004199
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase III Study of the Matrix Metalloprotease Inhibitor Prinomastat (AG3340) in Combination With Gemcitabine and Cisplatin in Patients Having Advanced Non-Small Cell Lung Cancer
Brief Title: Prinomastat and Combination Chemotherapy in Treating Patients With Metastatic or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AG-3340-017; CDR0000067442
Record Dates: First submitted 2000-01-21; First posted 2004-07-19 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; prinomastat

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: prinomastat

SUMMARY:
RATIONALE: Prinomastat may stop the growth of non-small cell lung cancer by stopping blood flow to the tumor. Drugs used in chemotherapy stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase III trial to determine the effectiveness of prinomastat plus cisplatin and gemcitabine in treating patients who have metastatic or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival, progression free survival, symptomatic progression free survival, and one year survival of patients with metastatic or recurrent non-small cell lung cancer treated with prinomastat (AG3340) or placebo in combination with gemcitabine and cisplatin. II. Compare the disease response and duration of response in these patients on these regimens. III. Compare the quality of life of these patients on these regimens. IV. Evaluate the safety of these regimens in these patients.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients receive oral prinomastat or placebo twice daily beginning on day 1, followed by gemcitabine IV on days 1 and 8 and cisplatin IV on day 1. Courses repeat every 3 weeks.

PROJECTED ACCRUAL: Approximately 420 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage IV or recurrent or T4 lesion non-small cell lung cancer Measurable or evaluable disease No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for non-small cell lung cancer Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Collier, Study Chair — Agouron Pharmaceuticals
Locations (1):
- Agouron Pharmaceuticals, Inc., La Jolla, California, United States